CLINICAL TRIAL: NCT05444595
Title: A Behavioral and Plant-Based Dietary Intervention to Improve Metabolic Health and Diabetes Risk Factors in an Underserved Latino Population
Brief Title: Behavioral Plant-Based Dietary Intervention in Latinos
Acronym: SB Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Sansum Diabetes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202308026
Record Dates: First submitted 2022-06-21; First posted 2022-07-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Metabolic Disease
Keywords: Latinos; Obesity; Plant-based diet
MeSH Terms: conditions — Obesity; Metabolic Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Behavioral and Plant-based Dietary Intervention (Experimental): In this arm, participants will receive the behavioral plant-based intervention from community health workers.
  Interventions: Behavioral: Behavioral plant-based dietary intervention
- Standard Care (Active Comparator): In this arm, participants will receive the standard care intervention from community health workers.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Behavioral plant-based dietary intervention — Participants will meet with community health workers to receive information focused on healthy eating and consuming a traditional plant-based diet in a group format for the first few months followed by individual check-ins.
  Arms: Behavioral and Plant-based Dietary Intervention
Behavioral: Standard care — Participants will meet with community health workers to receive general health information through individual check-ins.
  Arms: Standard Care

SUMMARY:
The Aims of this study are 1) to develop a traditional plant-based diet that is palatable and acceptable to the Latino population and which contains the appropriate calorie and macronutrient composition needed to lose weight and improve metabolic function and; 2) to develop a culturally sensitive [based on previous literature and stakeholder input] lifestyle intervention program, that will be delivered by community health workers [CHWs], that focuses on consuming a traditional plant-based diet and overcoming the barriers to incorporating this dietary therapy as part of the family lifestyle but with a focus on the adult participant with obesity. Ultimately, in Aim 3 the investigators will conduct a 16-week randomized controlled trial (RCT) in 40 Latino adults with obesity [20 control, 20 treatment] to evaluate the intervention's: i) clinical efficacy; ii) fidelity of the implementation by CHWs; and iii) acceptance by CHWs and study participants.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Hispanic and/or Latino heritage
* Body Mass Index (BMI) 30-42 kg/m²
* HbA1c ≤ 6.4%

Exclusion Criteria:

* Previous diagnosis of diabetes
* Unstable weight (≥4% during the last 2 months prior to study enrollment)
* Severe cardiovascular disease within the 6 months prior to study enrollment
* Severe organ system dysfunction
* active substance abuse with alcohol or drugs
* Severe anemia
* Pregnant or breastfeeding
* Use of medications that are known to affect the study outcome measures
* Persons who are not able to grant voluntary informed consent

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Body weight | Baseline and immediately after the intervention at 6 months
  Percent change in body weight from baseline to post-intervention

SECONDARY OUTCOMES:
Fat mass and fat free mass | Baseline and immediately after the intervention at 6 months
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
β-cell function | Baseline and immediately after the intervention at 6 months
  β-cell function will be assessed from a modified 3-hour oral glucose tolerance test
Insulin Clearance | Baseline and immediately after the intervention at 6 months
  Insulin clearance will be assessed from a modified 3-hour oral glucose tolerance test
Plasma Lipids | Baseline and immediately after the intervention at 6 months
  Fasting plasma lipid profile will be assessed by routine blood tests
Blood pressure | Baseline and immediately after the intervention at 6 months
  Systolic and diastolic blood pressure will be measured
Program acceptability from community health workers and study participants | Immediately after the intervention at 6 months
  Community health workers' and study participants' perceptions of program acceptability via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Jacome Sosa, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States